CLINICAL TRIAL: NCT02264171
Title: An Open Label Randomized Two-way Crossover Study to Investigate the Effect of Ketoconazole Mediated CYP3A4 Inhibition on the Single Oral Dose Pharmacokinetics of Tamsulosin in Healthy Male Volunteers (CYP2D6 Extensive Metabolizers)
Brief Title: Study to Investigate the Effect of Ketoconazole Mediated CYP3A4 Inhibition on Pharmacokinetics of Tamsulosin in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 527.78
Record Dates: First submitted 2014-10-14; First posted 2014-10-15 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — Tamsulosin; Ketoconazole

ARMS (2):
- Ketoconazole + Tamsulosin HCl (Experimental): Ketoconazole given once daily in the morning on days -3 to 2 Tamsulosin HCl given at day 1
  Interventions: Drug: Tamsulosin HCl; Drug: Ketoconazole
- Tamsulosin HCl (Active Comparator): Tamsulosin HCl given at day 1
  Interventions: Drug: Tamsulosin HCl

INTERVENTIONS:
Drug: Tamsulosin HCl
Drug: Ketoconazole
  Arms: Ketoconazole + Tamsulosin HCl

SUMMARY:
Study to investigate the effect of CYP3A4 inhibition by ketoconazole on the single oral dose pharmacokinetics of tamsulosin and to investigate the effect on safety and tolerability

ELIGIBILITY:
Inclusion Criteria:

All participants in the study will be

* Healthy males
* Ranging from 21 to 50 years of age
* Body mass index (BMI) within 18.5 to 29.9 kg/m2 (BMI calculation: weight in kilograms divided by the square of height in meters)
* In accordance with Good Clinical Practice (GCP) and the local legislation all volunteers will have given their written informed consent prior to admission to the study

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders, clinically relevant electrolyte disturbances
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of orthostatic hypotension, fainting spells or blackouts
* Chronic or clinically relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24:00 hours) within at least one month or less than ten half-lives of the respective drug before enrolment in the study or during the study
* Use of any drugs which might influence the results of the trial up to 7 days prior to enrolment in the study or during the study
* Participation in another trial with an investigational drug (within two months prior to administration or during the trial)
* Smoker (> 10 cigarettes or > 3 cigars of > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation (> 100 mL within four weeks prior to administration or during the trial)
* Any laboratory value outside the reference range if indicative of underlying disease or poor health
* Excessive physical activities within the last week before the trial or during the trial
* Hypersensitivity to treatment medication and/or related drugs of these classes
* Non extensive metabolizer (EM) for CYP2D6

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-04; Primary Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Cmax (maximum measured concentration of Tamsulosin HCl in plasma) | up to 48 hours after dosing
AUC0-∞ (Area under the concentration-time curve of Tamsulosin HCl in plasma over the time interval from 0 extrapolated to infinity) | up to 48 hours after dosing

SECONDARY OUTCOMES:
tmax (time from dosing to the maximum concentration of Tamsulosin HCl in plasma) | up to 48 hours after dosing
AUC0-tz (area under the concentration-time curve of Tamsulosin HCl in plasma over the time interval from 0 to the last quantifiable data point) | up to 48 hours after dosing
λz (terminal rate constant of Tamsulosin HCl in plasma) | up to 48 hours after dosing
t1/2 (terminal half-life of Tamsulosin HCl in plasma) | up to 48 hours after dosing
MRTpo (mean residence time Tamsulosin HCl in the body after oral administration) | up to 48 hours after dosing
CL/F (apparent clearance of the analyte in the plasma after extravascular administration) | up to 48 hours after dosing
Vz/F (apparent volume of distribution of Tamsulosin HCl during the terminal phase λz following an extravascular dose) | up to 48 hours after dosing
Number of subjects with adverse events | up to 21 days after last Tamsulosin administration
Assessment of tolerability by investigator on a 4-point scale | within 21 days after last Tamsulosin administration
Ratio of the Cmax value of the Test treatment to the Cmax value of the Reference treatment after single dose (RCmax,T/R) | up to 48 hours after dosing
Ratio of the Test treatment versus the Reference treatment from zero to infinity, expressed as ratio of AUC values after single dose (RAUC0-∞,T/R) | up to 48 hours after dosing